CLINICAL TRIAL: NCT05696483
Title: Phase 1 Randomized, Double-Blind, Single Ascending Dose, Multiple Ascending Dose, and Food Effect Study of the Safety, Tolerability, and Pharmacokinetics of OLX-07010 in Healthy Adult and Elderly Participants
Brief Title: Phase 1 Study of OLX-07010 in Healthy Adult and Elderly Participants
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Oligomerix, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OLX-07010-01
Record Dates: First submitted 2022-12-13; First posted 2023-01-25 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, four-part study of single ascending doses and multiple ascending doses in healthy adult participants, and as a single dose in healthy elderly participants. There is an option for an additional part to evaluate the effects of food.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: matching placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): Active OLX-07010 in single ascending and multiple ascending dose cohorts
  Interventions: Drug: OLX-07010 Active
- Placebo (Placebo Comparator): OLX-07010 placebo in single ascending and multiple ascending dose cohorts
  Interventions: Drug: OLX-07010 Placebo

INTERVENTIONS:
Drug: OLX-07010 Active — 25 and 75 mg capsules
  Arms: Active
Drug: OLX-07010 Placebo — 25 and 75 mg capsules
  Arms: Placebo

SUMMARY:
This First-in-human (FIH) study will evaluate the safety, tolerability, and pharmacokinetics of the tau self-association inhibitor, OLX-07010 in single ascending doses (SAD) and multiple ascending doses (MAD) in healthy adults (18-50 of age inclusive), and single dose in healthy elderly (51-75 of age inclusive). The effects of dosing with or without food in healthy adults will also be studied (optional).

DETAILED DESCRIPTION:
This FIH Phase 1 randomized, double-blind, four-part study will be conducted to evaluate the safety, tolerability, and PK of the tau self-association inhibitor, OLX-07010 in single ascending doses, multiple ascending doses in healthy adult participants, and as a single dose in healthy elderly participants. There is an option for an additional part to evaluate the effects of food (fed and fasted) on OLX-07010 in healthy adult participants. This study will be divided into 4 parts: Part 1-Randomized Double-Blind Single Ascending Dose in Healthy Adult Participants; Part 2-Randomized Double-Blind Multiple Ascending Dose in Healthy Adults Participants; Part 3-Randomized Double-Blind Single Dose in Healthy Elderly Participants; and Part 4 (Optional)-Food Effect (Single Cohort, 2 Sequence, 2 Period Crossover Fed and Fasted) in Healthy Adult Participants.

ELIGIBILITY:
Inclusion Criteria:

* Participant voluntarily agrees to participate and signs an approved informed consent prior to performing any of the Screening Visit procedures.
* Participant must be a healthy male or female of non-childbearing potential 18 to 50 years old inclusive, in Part 1, 2, and 4 of the study. Participant must be a healthy elderly male or female of non-childbearing potential 51-75 years old inclusive in Part 3 of the study.
* Male participants with body weight ≥ 55 kg; and females with body weight ≥ 50 kg and body mass index (BMI) between 18 and 30 kg/m2 (inclusive) for Part 1, 2, and 4 of the study; and BMI between 18 and 32 kg/m2 (inclusive) for Part 3 of the study.
* Female participants must be of non-childbearing potential (surgically sterile [hysterectomy or bilateral tubal ligation] or postmenopausal ≥ 1 year with follicle -stimulating hormone [FSH] > 40 IU/L at screening).

Exclusion Criteria:

* Participant has clinically significant history or evidence of cardiovascular (CV), respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or psychiatric disorder(s).
* Participant has any disorder that would interfere with the absorption, distribution, metabolism or excretion of drugs.
* Participant has a history of hypersensitivity to the study drug or any of the excipients or to medicinal products with similar chemical structures.
* Treatment with any investigational drug within the past 30 days prior to dosing.
* Use of any prescription drugs, herbal supplements, within 30 days prior to initial dosing, and over the counter (OTC) medication, dietary supplements (vitamins included) within 2 weeks prior to initial dosing. For elderly population in Part 3, allowed medications must be stable for at least 1 month.
* Clinically significant vital signs or ECG abnormality at screening and at baseline.
* Score of "yes" on specific items of the Suicidal Ideation section of the C-SSRS at the Screening Visit.
* History of any cancer within 5 years of screening (more than 10 years in remission).
* Any history of renal injury/kidney disease or presence of impaired renal function as indicated by clinically significantly abnormal creatinine or blood urea nitrogen (BUN) values in blood, or clinically relevant abnormal urinary constituents at Screening or Admission.
* Participant has any of the liver enzymes (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma glutamyl transferase [GGT]) or total bilirubin [TBL]) greater than the upper limit of normal (ULN), with the exception of isolated TBL elevation consistent with Gilbert's disease.
* Participants taking medications that are sensitive substrates for CYPC8, CYP2C19, CYP3A4, CYP1A2, and CYP2C9.
* Participant has a significant history of hypersensitivities or allergies to any medications, as determined by the PI/designee.
* Sexually active males not willing to use a condom during intercourse while taking the study drug and until EOS visit.
* Women of childbearing potential (WOCBP), defined as all women physiologically capable of becoming pregnant.
* Female participants are breastfeeding or female participants with a positive serum pregnancy test at the screening visit or positive urine pregnancy test at admission.
* Participants has poor venous access.
* Participant has history of alcohol and/or illicit drug abuse within 12 months prior dosing or positive alcohol/illicit drug test at screening and/or admission; smoking history (use of tobacco products in the previous 3 months prior dosing) or positive cotinine test at screening or admission.
* Participant has donated blood (> 500 mL) or blood products within 2 months prior to admission (Day -1). Plasma donation (> 200 mL) within 7 days prior to first dosing.
* Participant has previously been enrolled in this clinical study.
* Participant has a positive reverse transcription polymerase chain reaction (RT PCR) test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2).
* Participant has clinical signs and symptoms consistent with SARS-CoV-2 infection, e.g., fever, dry cough, dyspnea, sore throat, fatigue, or laboratory confirmed acute infection with SARS-CoV-2.
* Participant who had a severe course of COVID-19; (extracorporeal membrane oxygenation, mechanically ventilated, or Intensive Care Unit stay).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2023-01-20 (Actual); Primary Completion 2026-01-02 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as Measured by NCI-CTCAE criteria | After each dose of OLX-07010 through completion of dosing, up to 30 days
  Safety and tolerability of OLX-07010 will be assessed by documenting adverse events occurring after single dose administration (Parts 1, 3 and 4) and multiple dose administration (Part 2)
Incidence of Treatment-Emergent Adverse Events as Measured by Clinical Laboratory Measurements According to Established Clinical Normal Ranges | Change from baseline at 2-4 hours post-dose of OLX-07010
  Blood and Urine samples will be taken after administration of OLX-07010 and values will be compared to baseline and established normal ranges to determine how OLX-07010 administration impacts normal body function
Incidence of Treatment-Emergent Adverse Events as Measured by ECG | Change from baseline at 2, 4, and 8 hours and Days 2 and 4 post-dose of OLX-07010
  ECGs will be used to measure changes to the heart after administration of OLX-07010
Incidence of Treatment-Emergent Adverse Events as Measured by Neurological Examination | Change from baseline at Day 1, Day 4 (Parts 1 and 3) and Days 7 and 10 (Parts 2 and 4) post-dose of OLX-07010
  Neurological assessments will be performed to investigate the potential effect of the study drug on mental status, gait (normal/abnormal), coordination/incoordination, tremor, muscle tone, stereotypy and biceps reflexes

SECONDARY OUTCOMES:
Maximum drug concentration in plasma (Cmax) of OLX-07010 after single ascending doses | Blood collection on Day 1, 2, 3, and 4. On Day 1 (pre-dose 0 hour, post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, 7, 9, and 12 hours), Day 2 (24 hours post-dose), Day 3 (48 hours post-dose) and Day 4 (72 hours post-dose).
  The maximum drug concentration will be determined after a single ascending doses
Maximum drug concentration in plasma (Cmax) of OLX-07010 after multiple ascending doses | Day 1and Day 7 (pre-dose 0 hour, and post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, 7, 9, 12 hours), Days 2 (24 hours post-dose) to Day 6 (pre-dose 0 hours), Day (24 hours post-dose), Day 9 (48 hours post-dose), and Day 10 (72 hours post-dose).
  The maximum drug concentration will be determined after a single ascending doses
Area under the concentration-time curve in plasma (AUC) of OLX-07010 after single ascending doses. | Blood collection on Day 1, 2, 3, and 4. On Day 1 (pre dose 0 hour, post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, 7, 9, and 12 hours), Day 2 (24 hours post-dose), Day 3 (48 hours post-dose) and Day 4 (72 hours post-dose).
  Determine the Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration (tlast) and from pre-dose (time 0) extrapolated to infinite time (AUClast + Clast/λz) calculated using the linear-log trapezoidal rule.
Area under the concentration-time curve in plasma (AUC) of OLX-07010 after multiple ascending doses. | Day 1and Day 7 (pre-dose 0 hour, and post-dose at 15 minutes, 30 minutes, 1, 1.5, 2, 3, 4, 5, 7, 9, 12 hours), Days 2 (24 hours post-dose) to Day 6 (pre-dose 0 hours), Day (24 hours post-dose), Day 9 (48 hours post-dose), and Day 10 (72 hours post-dose).
  Determine the Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration (tlast) and from pre-dose (time 0) extrapolated to infinite time (AUClast + Clast/λz) calculated using the linear-log trapezoidal rule.
Renal clearance and percent drug excreted in Urine after single and multiple ascending doses of OLX-07010. | Part 1:Day 1 at 0 hour (pre-dose), 0-4; 4-8; 8-12; and 12-24 hours post-dose. Part 2: Day 1 and Day 7 at 0 hour (pre-dose), 0-4 hours; 4-8 hours; 8-12 hours; 12-24 hours.
  Determine the the renal clearance and amount of OLX-07010 excreted in urine.

CONTACTS AND LOCATIONS:
Locations (1):
- California Clinical Trials Medical Group, Inc, Glendale, California, United States

IPD SHARING:
Plan to Share IPD: No